CLINICAL TRIAL: NCT03909217
Title: Effectiveness and Safety of Transcutaneous Electrical Cranial-auricular Acupoint Stimulation (TECAS) for Patients With Mild-to-moderate Depression.
Brief Title: Treating Depression With Transcutaneous Electrical Cranial-auricular Acupoint Stimulation (TECAS).
Acronym: TECAS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Beijing First Hospital of integrated Chinese and Western Medicine (Other); The First Hospital of Hebei Medical University (Other); Southwest Medical University (Other)
Responsible Party: Principal Investigator, Prof. Zhang Zhang-Jin, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018YFC1705801
Record Dates: First submitted 2019-03-28; First posted 2019-04-09 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Mild-to-moderate Depression
Keywords: Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TECAS (Experimental): Patients will receive transcutaneous electrical cranial-auricular acupoint stimulation (TECAS) daily.
  Interventions: Procedure: TECAS Procedure; Drug: Insomnia medication
- Anti-depressants (Active Comparator): Each subject shall receive oral administration Escitalopram (10-20mg/day, q.d.), as prescribed by a clinical psychiatrist with respect to patients' conditions for 8 consecutive weeks.
  Interventions: Drug: Escitalopram; Drug: Insomnia medication

INTERVENTIONS:
Procedure: TECAS Procedure — Location:
  1. Cranial electrical stimulation acupoints: Baihui (DU20) and Yintang (DU29).
  2. Auricular electrical stimulation zone: the distribution area of auricular branch of the vagus nerve.
  Two electrodes electric stimulation at a frequency of 4/20 Hz will be employed on the cranial acupoints and the auricular zone respectively. The TECAS treatment will consistent of two sessions per day (30 minutes) for 8 consecutive weeks.
  Other Names: TECAS
  Arms: TECAS
Drug: Escitalopram — Each subject shall receive oral administration Escitalopram (10-20mg/day, q.d.), as prescribed by clinical psychiatrist with respect to patients' conditions for 8 consecutive weeks.
  Other Names: Escitalopram Oxalate Tablets
  Arms: Anti-depressants
Drug: Insomnia medication — For patients with severe insomnia, stabilizers and benzodiazepines could be prescribed and must be recorded in the case report form.
  Other Names: Benzo

SUMMARY:
One multi-center, randomized controlled clinical trial is designed to examine whether transcutaneous electrical cranial-auricular acupoint stimulation (TECAS) is non-inferior to the antidepressant drug (Escitalopram) in treating mild-to-moderate depression, to evaluate the depressive subtypes who are suitable for the TECAS treatment. To achieve this objective, 470 patients with mild-to-moderate depression will be recruited and assigned to receive TECAS treatment (n =235) or Escitalopram (n =235, 10-20mg/day, q.d.) for 8 weeks. The primary outcome is the Montgomery-Åsberg Depression Rating Scale (MADRS); other outcomes include the17-item Hamilton Depression Scale (HAMD-17), the Hamilton Anxiety Rating Scale (HAMA), Pittsburgh sleep quality index (PSQI), the Short Form 36 Health Survey and TCM diagnosis of depression. In addition, the safety index will be measured throughout the whole study.

DETAILED DESCRIPTION:
Depression is a common and costly disorder with high prevalence rate and high suicide rate. Antidepressants are the first-line treatments for depression. However, approximately 50% to 60% of the patients have not achieved adequate response following antidepressant treatment.

A large body of evidence well confirms that electro-acupuncture is effective in improving depression and reducing anti-depressant treatment-caused side effects, including pain, nausea, dizziness, fatigue, anxiety and sleep disturbance.

Based on the combination of ancient and modern literature and famous traditional Chinese medicine practitioners' experience, the Evidence-based Guidelines of Clinical Practice with Acupuncture and Moxibustion-Depression (ZJ/TE003-2014) recommended Baihui (DU20) and Yintang (DU29) as main acupoints in treating patients with depression via electro-acupuncture.

Our research team have completed a series of clinical trials, including electrical stimulation on cranial and auricular acupoints for treating depression, postpartum depression, post-stroke depression, and depression with somatic pain. These studies found that cranial-auricular acupoint stimulation, as well as transcutaneous electrical stimulation, can improve depressive symptoms and accompanying symptoms in patients with depression significantly.

Unlike traditional acupuncture, transcutaneous electrical stimulation does not need needles to penetrate the skin. It places electrodes on the skin of the corresponding acupoints. In this way, traumatic pain and fear of acupuncture can be avoided. And it is more easily accepted for patients and more convenient for clinical operation. Therefore, the investigators plan to build a novel transcutaneous electrical stimulation therapy--Transcutaneous electrical cranial-auricular acupoint stimulation (TECAS).

In the proposed study, a combination of transcutaneous electrical cranial and transcutaneous electrical auricular acupoint stimulation will be employed to treat patients with mild-to-moderate depression compared with antidepressant Escitalopram, to confirm the clinical effectiveness of TECAS in mild-to-moderate depression.

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis as mild to moderate depression；
2. Aged 18-70；
3. A score of MADRS ≥12 and <30 without suicide risk;
4. Participants to give consent and to cooperate with the treatment and data collection;

Exclusion Criteria:

1. Pregnant；
2. Patients with severe diseases of heart, brain, liver, kidney or hematopoietic system, patients with acute diseases, infectious diseases and malignant tumours;
3. Patients who are unable to stop taking relevant drugs as required during the trial; (any other drug or non-drug treatment that affects depressive symptoms, including Chinese medicine, western medicine, and physical therapies et al.)
4. Patients with any history of psychosis or mania;
5. Patients with cognitive disorders or personality disorders;
6. Patients with serious suicidal ideation or behaviours.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Clinical response at the end of treatment | 8 week
  The responder is defined as a ≥50% reduction from the baseline MADRS or HAMD-17 at the end of treatment.

SECONDARY OUTCOMES:
Remission at the end of treatment | 8 week
  Remission is defined as a score of 12 or fewer points on the MADRS or as 7 or fewer points on the HAMD-17.
Changes from baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) score | Baseline, 2 week, 4 week, 8 week, 12 week
  The 10-item Montgomery-Åsberg Depression Rating Scale (MADRS) measures severity of depression in individuals 18 years and older (range, 0 to 60, with higher scores indicating more severe depression; minimal clinically significant difference, 1.6 to 1.9 points). Each item is rated on a 7-point scale. The scale is an adaptation of the Hamilton Depression Rating Scale and has a greater sensitivity to change over time. The scale takes 20 to 30 minutes to complete and score.
Changes from baseline in the 17-item Hamilton Depression Scale (HAMD-17) | Baseline, 2 week, 4 week, 8 week, 12 week
  The Hamilton Rating Scale for Depression, abbreviated HDRS, HRSD or HAM-D, measures depression in individuals before, during and after treatment. The scale is administered by a health care professionals and contains 21 items, but is scored based on the first 17 items, which are measured either on 5-point or 3-point scales. It takes 15 to 20 minutes to complete and score.
Changes from baseline in the Hamilton Anxiety Rating Scale (HAMA) | Baseline, 2 week, 4 week, 8 week, 12 week
  The HAMA is widely used in both clinical practice and research settings. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Changes from baseline in the Pittsburgh sleep quality index (PSQI) | Baseline, 2 week, 4 week, 8 week, 12 week
  The sleep quality will be assessed using the Pittsburgh sleep quality index. Assessments will be conducted at baseline, 2-week and once every four weeks thereafter.
Changes from baseline in the Short Form 36 Health Survey | Baseline, 2 week, 4 week, 8 week, 12 week
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. It has 36 items grouped in 8 dimensions: physical functoning, physicial and emotional limitations, social functioning, bodily pain, general and mental health.
Adverse events | Weeks 1-12
  Adverse events of TECAS treatment will be assessed and would be evaluated during the whole procedure, as well as laboratory tests (whole blood counts, renal and liver functions) if needed. Side Effects of Escitalopram will be assessed and would be evaluated during the whole procedure, as well as laboratory tests (whole blood counts, renal and liver functions) if needed. All clinical adverse events will be recorded in terms of intensity (mild, moderate, or severe), duration, outcome and relationship to the study.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang-Jin ZHANG, BMed, PhD, Principal Investigator — School of Chinese Medicine, The University of Hong Kong
Locations (6):
- China (6):
  - Department of Chinese Medicine, The University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - Department of neurology, The University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - The First Hospital of Hebei Medical University, Hebei, Shijiazhuang
  - Southwest Medical University, Hospital of Traditional Chinese Medicine, Luzhou, Sichuan
  - Beijing First Hospital of Integrated Chinese and Western Medicine, Beijing
  - Guang'anmen Hospital of the Chinese Academy of Chinese Medical Science, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong YK, Wu JM, Zhou G, Zhu F, Zhang Q, Yang XJ, Qin Z, Zhao N, Chen H, Zhang ZJ. Antidepressant Monotherapy and Combination Therapy with Acupuncture in Depressed Patients: A Resting-State Functional Near-Infrared Spectroscopy (fNIRS) Study. Neurotherapeutics. 2021 Oct;18(4):2651-2663. doi: 10.1007/s13311-021-01098-3. Epub 2021 Aug 24. PMID 34431029
- [Background] Zhang ZJ, Man SC, Yam LL, Yiu CY, Leung RC, Qin ZS, Chan KS, Lee VHF, Kwong A, Yeung WF, So WKW, Ho LM, Dong YY. Electroacupuncture trigeminal nerve stimulation plus body acupuncture for chemotherapy-induced cognitive impairment in breast cancer patients: An assessor-participant blinded, randomized controlled trial. Brain Behav Immun. 2020 Aug;88:88-96. doi: 10.1016/j.bbi.2020.04.035. Epub 2020 Apr 16. PMID 32305573
- [Background] Zhang ZJ, Zhao H, Jin GX, Man SC, Wang YS, Wang Y, Wang HR, Li MH, Yam LL, Qin ZS, Yu KT, Wu J, Ng FB, Ziea TE, Rong PJ. Assessor- and participant-blinded, randomized controlled trial of dense cranial electroacupuncture stimulation plus body acupuncture for neuropsychiatric sequelae of stroke. Psychiatry Clin Neurosci. 2020 Mar;74(3):183-190. doi: 10.1111/pcn.12959. Epub 2019 Dec 20. PMID 31747095
- [Background] Fang J, Rong P, Hong Y, Fan Y, Liu J, Wang H, Zhang G, Chen X, Shi S, Wang L, Liu R, Hwang J, Li Z, Tao J, Wang Y, Zhu B, Kong J. Transcutaneous Vagus Nerve Stimulation Modulates Default Mode Network in Major Depressive Disorder. Biol Psychiatry. 2016 Feb 15;79(4):266-73. doi: 10.1016/j.biopsych.2015.03.025. Epub 2015 Apr 2. PMID 25963932
- [Background] Tu Y, Fang J, Cao J, Wang Z, Park J, Jorgenson K, Lang C, Liu J, Zhang G, Zhao Y, Zhu B, Rong P, Kong J. A distinct biomarker of continuous transcutaneous vagus nerve stimulation treatment in major depressive disorder. Brain Stimul. 2018 May-Jun;11(3):501-508. doi: 10.1016/j.brs.2018.01.006. Epub 2018 Jan 31. PMID 29398576
- [Derived] Yang S, Qin Z, Yang X, Chan MY, Zhang S, Rong P, Hou X, Jin G, Xu F, Liu Y, Zhang ZJ. Transcutaneous Electrical Cranial-Auricular Acupoint Stimulation vs. Escitalopram for Patients With Mild-to-Moderate Depression (TECAS): Study Design for a Randomized Controlled, Non-inferiority Trial. Front Psychiatry. 2022 May 10;13:829932. doi: 10.3389/fpsyt.2022.829932. eCollection 2022. PMID 35619617